CLINICAL TRIAL: NCT00141232
Title: A Multicentre, Randomised, Double Blind Placebo Controlled Trial Evaluating Atorvastatin in Factorial With Omega-3 Fatty Acids Cardiovascular Risk Reduction in Patients With Type 2 Diabetes
Brief Title: Evaluating Atorvastatin With Omega-3 Fatty Acids in Cardiovascular Risk Reduction in Patients With Type 2 Diabetes
Acronym: AFORRD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: Churchill Hospital (Other)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: A2581114
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Atorvastatin; Fatty Acids, Omega-3

INTERVENTIONS:
Drug: Atorvastatin and Omega-3 fatty acids

SUMMARY:
The AFORRD trial is asking three important questions:

What proportion of people with Type 2 Diabetes are likely to be treated satisfactorily with a fixed dose of a statin that lowers blood cholesterol levels to help reduce the risk of heart disease? To what extent do omega-3 fatty acids lower blood triglyceride levels when given with or without a statin? Are there simple techniques that can help people to take their tablets on a regular basis?

ELIGIBILITY:
Inclusion Criteria:

* They have a diagnosis of Type 2 Diabetes Mellitus for at least 3 months prior to entry.
* Are not known to have had a cardiovascular event

Exclusion Criteria:

* They are taking prescribed lipid lowering therapy
* Have triglycerides > or = 8.0 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2004-11; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Prim objective (16 wks) for atorvastatin: Proportion of pats. who achieve measured
LDL levels <2.6 mmol/L (<100 mg/dl) Prim object (16 wks) for Omega-3 fatty acid:
Prop of pats. who achieve measured triglycerides <1.5 mmol/L (<200 mg/dl)

SECONDARY OUTCOMES:
Prop of pats who achieve LDL levels <2.6 mmol/L (<100 mg/dl) at 52 weeks, taking into account whether the patient received additional atorvastatin therapy or placebo at week 16.
Prop of pats who achieve triglycerides <1.5 mmol/L (<200 mg/dl) at 52 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United Kingdom (52):
  - Pfizer Investigational Site, Irvine, Ayrshire
  - Pfizer Investigational Site, Farnworth, Bolton
  - Pfizer Investigational Site, Thornhill, Cardiff
  - Pfizer Investigational Site, Fowey, Cornwall
  - Pfizer Investigational Site, Launceston, Cornwall
  - Pfizer Investigational Site, Penzance, Cornwall
  - Pfizer Investigational Site, Saltash, Cornwall
  - Pfizer Investigational Site, St Austell, Cornwall
  - Pfizer Investigational Site, Darlington, County Durham
  - Pfizer Investigational Site, Newton Aycliffe, County Durham
  - Pfizer Investigational Site, Three Bridges, Crawley
  - Pfizer Investigational Site, Plymouth, Devon
  - Pfizer Investigational Site, Bexhill-on-Sea, East Sussex
  - Pfizer Investigational Site, Bath, England
  - Pfizer Investigational Site, Dronfield, Sheffield, England
  - Pfizer Investigational Site, Surrey, England
  - Pfizer Investigational Site, Halstead, Essex
  - Pfizer Investigational Site, Stonehouse, Gloucestershire
  - Pfizer Investigational Site, Southampton, Hampshire
  - Pfizer Investigational Site, Hildenborough, Kent
  - Pfizer Investigational Site, Thorneton-Clevely, Lancashire
  - Pfizer Investigational Site, Balham, London
  - Pfizer Investigational Site, Fulham, London
  - Pfizer Investigational Site, Tooting, London
  - Pfizer Investigational Site, Hayes, Middlesex
  - Pfizer Investigational Site, Wellingborough, Northamptonshire
  - Pfizer Investigational Site, Cookstown, Northern Ireland
  - Pfizer Investigational Site, Frome, Somerset
  - Pfizer Investigational Site, Fetcham, Surrey
  - Pfizer Investigational Site, Woking, Surrey
  - Pfizer Investigational Site, Crawley, West Sussex
  - Pfizer Investigational Site, Leeds, West Yorkshire
  - Pfizer Investigational Site, Bradford-on-Avon, Wiltshire
  - Pfizer Investigational Site, Melksham, Wiltshire
  - Pfizer Investigational Site, Swindon, Wiltshire
  - Pfizer Investigational Site, Trowbridge, Wiltshire
  - Pfizer Investigational Site, Warminster, Wiltshire
  - Pfizer Investigational Site, Sheffield, Yorkshire
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Belfast
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Bucks
  - Pfizer Investigational Site, Chesterfield
  - Pfizer Investigational Site, Chippenham, Wiltshire
  - Pfizer Investigational Site, Cornwall
  - Pfizer Investigational Site, County Antrim, Northern Ireland
  - Pfizer Investigational Site, Darlington
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, East Sussex
  - Pfizer Investigational Site, Isle of Wight
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Westbury

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581114&StudyName=Evaluating+Atorvastatin+with+Omega%2D3+Fatty+Acids+in+Cardiovascular+Risk+Reduction+in+Patients+with+Type+2+Diabetes